CLINICAL TRIAL: NCT06484712
Title: The Role of Sensory Deficits in the Neural Control of Balance During Walking in People With Functional Ankle Instability
Brief Title: Electrical Stimulation Effect on Ankle Instability During Walking in Virtual Reality Setup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2182823-1
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-06

CONDITIONS: Ankle Sprains; Ankle Instability
Keywords: Chronic Ankle Instability; Electrical Stimulation; Virtual Reality; Balance; Locomotor Control
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Cross sectional study of responses to visual perturbations in one group, people with chronic ankle instability. Each participant will undergo two stimulation conditions, stochastic resonance (SR) stimulation and a control / no stochastic resonance (no-SR) condition while walking with and without visual perturbations.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stochastic Resonance (SR) (Experimental): During this condition, participants will walk on the treadmill while receiving SR stimulation at their individual optimal intensity (SR) with and without visual perturbations.
  Interventions: Device: Stochastic Resonance (SR)
- No Stochastic Resonance (no-SR) (No Intervention): During this condition, participants will walk on the treadmill while receiving no SR stimulation (no-SR) with and without visual perturbations.

INTERVENTIONS:
Device: Stochastic Resonance (SR) — The system consists of six linear isolated stimulators (STMISOLA, Biopac Systems, Inc., Goleta, USA). The SR signal (Gaussian White Noise, zero mean) will be generated through a 16 bit PCI 6733 National Instruments multifunction data acquisition card by a custom LabView program. The stimulation sites include the ankle, lateral soleus, peroneus longus, and tibialis anterior muscles and the hip.
  Arms: Stochastic Resonance (SR)

SUMMARY:
The purpose of the study is to investigate whether electrical stimulation to leg muscles and joints can help with balance in people with ankle instability. Participants will be asked to walk on a treadmill in a virtual reality cave. They will receive light electrical stimulation at the legs to improve your balance. The virtual reality image will sometimes shift in unexpected ways to challenge your balance. During the session, we will conduct a series of clinical assessments, including tests of functional performance and balance. Additionally, participants will be asked to fill out some questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 39 years.
* Having at least one significant ankle sprain in the past year, which causes a minimum of one interrupted day of physical activity.
* Having a history of at least two ankle sprains or "giving way" sensations at the injured ankle and/or a history of general feeling of ankle joint instability associated with the fear of getting another acute ankle sprain.
* Score < 24 in the Cumberland Ankle Instability Tool (CAIT), and/or > 11 in the Identification of Functional Ankle Instability (IdFAI), and/or answer ''yes'' to at least 5 yes/no questions in the Ankle Instability Instrument (AII).

Exclusion Criteria:

* Any head, neck, or face injury in the six months prior to the study (e.g., concussion, eye injury).
* History of vestibular or ocular dysfunction.
* Currently taking any medications affecting balance (i.e. antibiotics).
* History of injuries to lower extremities including fractures, knee injuries, and hip injuries.
* Sustaining an ankle sprain injury in the last 6 weeks.
* Pregnancy
* Any neurological disorders (e.g., seizure disorders, closed head injuries with loss of consciousness greater than 15 minutes, CNS neoplasm, history of stroke)
* Unstable cardiac or pulmonary disease.
* Clinically obese (BMI 30 or above).
* Any metal implant in the feet or legs that is close to the stimulating electrodes.
* A known allergy to medical-grade adhesives.
* Any other comorbidity affecting the ability to safely walk without assistance for at least 2 minutes

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Change in the Center of Mass (CoM) excursion | At the end of the session after 12 walking trials of randomized stimulation.
  For the visual perturbation trials, we will use CoM excursion as the primary outcome measure since it has been used in prior studies in children and adults using visual perturbation protocols. This is determined by comparing the average CoM during perturbed steps to non-perturbed steps for each participant, integrated across the first eight steps initiated by the heel strike that triggered the stimulus. We will measure CoM using kinetics and kinematic computed through a motion capture system(Qualysis).
  For the unperturbed trials, we will use margin of stability (MoS) as the primary outcome measure. MOS refers to the distance between extrapolated center of mass, which includes center of mass position and velocity, and the base of support. It has been previously used to measure balance in children with cerebral palsy and Parkinson Disease.

CONTACTS AND LOCATIONS:
Overall Officials: John Jeka, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided